CLINICAL TRIAL: NCT04631068
Title: A Prospective, Randomized, Multicentric Clinical Evaluation Comparing a Monofocal Extended Depth of Focus IOL With a Monofocal IOL
Brief Title: Clinical Comparison of a Monofocal eDOF IOL With a Monofocal IOL
Acronym: MonoeDOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Vision Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVS CP-7944
Record Dates: First submitted 2019-10-22; First posted 2020-11-17 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Patients participating will be randomised to either receive the Mono-EDoF ME4 Intraocular Lens (IOL) in both eyes or the TECNIS ZCB00 IOL in both eyes. Twice as many subjects will receive the Mono-EDoF ME4 IOL compared to the TECNIS ZCB00 IOL.
  Both IOLs have received the CE marked. The aim with both IOLs is to provide patients good vision at distance with no glasses. The Mono-eDoF ME4 might offer the additional benefit of achieving good vision at intermediate distance without glasses.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Santen xact Mono-EDoF ME4 Intraocular Lens (IOL) (Active Comparator): The Monofocal Extended Depth of Focus (Mono-EDoF) posterior chamber foldable intraocular lens is ultraviolet and blue-light absorbing designed to be positioned in the lens capsule to replace the optical function of the natural crystalline lens. The diffractive technology of the IOL allows most of the light to converge in one focal point thereby providing high quality of distance vision and continuous focus to intermediate vision while minimizing the effects of unwanted visual disturbances. The visual quality is expected to be similar to monofocal IOLs.
  Surgery to implant the Mono-EDoF ME4 Intraocular Lens (IOL) will be performed on Day 0 of the study, using standard microsurgical techniques. All instruments and procedures used will be identical to those routinely used for small incision phacoemulsification.
  Interventions: Procedure: Cataract surgery
- J&J TECNIS ZCB00 Intraocular Lens (IOL) (Placebo Comparator): The TECNIS 1-Piece Intraocular Lens (IOL), Model ZCB00, is a standard monofocal ultraviolet light absorbing posterior chamber IOL, which is designed to be positioned in the lens capsule to replace the optical function of the natural crystalline lens.
  Surgery to implant the TECNIS ZCB00 Intraocular Lens (IOL) will be performed on Day 0 of the study, using standard microsurgical techniques. All instruments and procedures used will be identical to those routinely used for small incision phacoemulsification.
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Small incision cataract surgery with implantation of an intraocular lens

SUMMARY:
Post-market, prospective, randomized, single-masked, multi-center clinical study investigating the safety and effectiveness of the Monofocal Extended Depth of Focus Intraocular Lens (Mono-EDoF IOL) when compared to a Standard Monofocal Intraocular Lens.

Primary Objectives:

* To evaluate the distance VA of the study IOLs
* To evaluate the intermediate VA of the study IOLs
* To explore the safety profile with regards to visual disturbances

DETAILED DESCRIPTION:
This study is aimed at patients who have a cloudy lens in both of their eyes, and are eligible for cataract surgery with implantation of an intraocular lens. Patients should be otherwise healthy with no other eye diseases.

The study will take place in 3 centers in Europe, including Oxford Eye Hospital, a part of Oxford University Hospitals NHS Trust and will include 70 patients in total.

The aim of the study is to investigate the safety and effectiveness of a new Intraocular Lens (IOL): the Monofocal Extended Depth of Focus (Mono-EDoF ME4) IOL and to compare it to a standard Monofocal IOL (TECNIS ZBC00). Patients participating will be randomised to either receive the Mono-EDoF ME4 IOL in both eyes or the TECNIS ZCB00 IOL in both eyes. Twice as many subjects will receive the Mono-EDoF ME4 IOL compared to the TECNIS ZCB00 IOL.

Both IOLs have received the CE marked. The aim with both IOLs is to provide patients good vision at distance with no glasses. The Mono-eDoF ME4 might offer the additional benefit of achieving good vision at intermediate distance without glasses.

Total duration of clinical investigation is 12 months and the total expected duration for each patient is 8 months.

Patients will be screened for eligibility preoperatively obtaining a medical history and to establish a baseline ocular condition. Surgeries will be performed on different dates for both eyes but not more than one month apart. The patient will need to return to for seven follow-up visits after eye surgery where vision and health of the eye will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 22 years of age and older at the time of consent.
2. Cataracts in both eyes.
3. Expected post-operative refractive astigmatism of ≤ 1.0 D.
4. Calculated lens power from 18 D to 30 D for both study IOLs.
5. Willing and able to return for all scheduled treatment and post-operative visits for a minimum of 6 months.
6. Planned removal of visually significant cataract (cortical, nuclear, posterior subcapsular, or a combination) by phacoemulsification cataract extraction in both eyes.
7. Willing to discontinue contact lens wear, if applicable, and demonstrate corneal stability prior to biometry and surgery.
8. Preoperative best corrected distance visual acuity (BCDVA) of 20/32 or worse, with or without a glare source, or preoperative BCDVA of 20/25 or worse with patient complaining of severe visual disturbances attributable to cataract.
9. Post-operative BCVA projected to be 0.2 LogMAR or better (as determined by the medical judgment of the Investigator or measured by potential acuity meter / retinal acuity meter (PAM / RAM) if necessary).
10. Pharmacologically dilated pupil size at least 6.0 mm.
11. Must be able to understand and provide informed consent themselves or through a representative with a witness present on the IRB or EC approved Informed Consent Form (ICF).

Exclusion Criteria:

1. Participation in any other drug or device clinical trial within 30 days prior to enrolling in this study and/or during study participation.
2. Pregnancy or lactation.
3. Subject who, in the clinical judgment of the Investigator, is not suitable for participation in the study for another clinical reason, as documented by the investigator (reason to be documented by the site on Case Report Forms - CRF's).
4. Any type of cataract (e.g., traumatic, congenital, polar) other than those noted in inclusion criteria.
5. History of any intraocular or corneal surgery in either eye (including LASIK, PRK, etc.).
6. Ocular conditions which could affect the stability of the IOL (e.g., pseudoexfoliation, zonular dialysis, evident zonular weakness or dehiscence, etc.) in either eye.
7. Any anterior segment pathology likely to increase the risk of complications from phacoemulsification cataract extraction (e.g., chronic uveitis, iritis, iridocyclitis, aniridia, rubeosis iridis, clinically significant corneal disease, Fuchs, or anterior membrane dystrophies, etc.) in either eye.
8. Mature cataract that is likely to prolong phacoemulsification and/or lead to intraoperative complications prior to attempted IOL implantation.
9. Any visually significant intraocular media opacity other than cataract in either eye.
10. History of any clinically significant retinal pathology or ocular diagnosis (e.g., diabetic retinopathy, ischemic disease, macular degeneration, retinal detachment, amblyopia, optic neuropathy, microphthalmos, aniridia, etc.) in either eye that could alter or limit final postoperative visual prognosis.
11. History of cystoid macular edema in either eye.
12. Severe dry eye that, in the opinion of the investigator, would impair the ability to obtain reliable study measurements.
13. Uncontrolled (e.g., non-medicated) glaucoma in either eye.
14. Extremely shallow anterior chamber (< 2.0 mm).
15. Subjects with large refractive errors (hyperopia/myopia) of axial or pathologic origin that, in the opinion of the investigator, could confound outcomes.
16. Irregular astigmatism, corneal degeneration or dystrophy.
17. Uncontrolled systemic disease (e.g., diabetes mellitus, active cancer treatment, mental illness, etc.) in the opinion of the Investigator, would put the subject's health at risk and/or prevent the subject from completing all study visits.
18. Systemic medication that, in the opinion of the investigator, may confound the outcome or increase the intraoperative and post-operative risk to the subject (e.g., Tamsulosin Hydrochloride) or other medications including anticholinergics, alpha adrenergic blocking agents with similar side effects (e.g., small pupil/floppy iris syndrome).
19. Subjects who may reasonably be expected to require any additional ophthalmic surgical intervention at any time during the study (other than YAG capsulotomy).
20. Need for concomitant procedures (e.g., glaucoma surgery, RK, LASIK, etc.).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Monocular Uncorrected Distance VA at Visit 4 (Month 3) | 80-100 days after second eye surgery
  Monocular uncorrected distance visual acuity measured using ETDRS visual acuity chart

SECONDARY OUTCOMES:
Monocular Distance Corrected Intermediate VA at Visit 4 (Month 3) | 80-100 days after second eye surgery
  Subject's vision is corrected for distance and then subject's intermediate vision is measured using a 66-cm ETDRS chart.
Monocular Uncorrected Intermediate VA at Visit 4 (Month 3) | 80-100 days after second eye surgery
  Intermediate Visual Acuity is measured using a 66-cm ETDRS chart.

OTHER OUTCOMES:
Safety endpoints | Baseline, Day 0 (Surgery), Visit 1 (Day 1), Visit 2 (Week 1), Visit 3 (Month 1), Visit 4 (Month 3), and Visit 5 (Month 6)
  The primary safety endpoint is the overall safety profile of the study IOLs as reflected by rates of adverse events.
Safety endpoints | Baseline, Visit 3 (Month 1), Visit 4 (Month 3), and Visit 5 (Month 6)
  The primary safety endpoint is the overall safety profile of the study IOLs as reflected by loss of BCDVA.
Safety endpoints | Baseline, Visit 1 (Day 1), Visit 2 (Week 1), Visit 3 (Month 1), Visit 4 (Month 3), and Visit 5 (Month 6)
  The primary safety endpoint is the overall safety profile of the study IOLs as reflected by slit lamp examination.
Safety endpoints | Baseline, Visit 5 (Month 6)
  The primary safety endpoint is the overall safety profile of the study IOLs as reflected by dilated fundus exam.
Safety endpoints | Baseline, Visit 1 (Day 1), Visit 2 (Week 1), Visit 3 (Month 1), Visit 4 (Month 3), and Visit 5 (Month 6)
  The primary safety endpoint is the overall safety profile of the study IOLs as reflected by intraocular pressure.
Safety endpoints | Day 0 (Surgery), Visit 1 (Day 1), Visit 2 (Week 1), Visit 3 (Month 1), Visit 4 (Month 3), and Visit 5 (Month 6)
  The primary safety endpoint is the overall safety profile of the study IOLs as reflected by device deficiencies.
Safety endpoints | Baseline, Day 0 (Surgery), Visit 1 (Day 1), Visit 2 (Week 1), Visit 3 (Month 1), Visit 4 (Month 3), and Visit 5 (Month 6)
  The primary safety endpoint is the overall safety profile of the study IOLs as reflected by visual symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, MD, Study Chair — Medical Monitor
Locations (3):
- University Hospital Pellegrin, Bordeaux, Cedex, France
- Hospital de Braga, Braga, Portugal
- Oxford Eye Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Black S. Successful Restoration of Visual Acuity with an Extended Range of Vision Intraocular Lens after Multifocal Laser Ablation. Case Rep Ophthalmol. 2016 Oct 11;7(3):193-197. doi: 10.1159/000450675. eCollection 2016 Sep-Dec. PMID 28101037
- [Background] Bostanci Ceran B, Takmaz T, Can I, Demirok G, Uysal BS. Clinical outcomes and optical performance of four differentmultifocal intraocular lenses. Turk J Med Sci. 2016 Apr 19;46(3):597-603. doi: 10.3906/sag-1403-24. PMID 27513232
- [Background] Cillino S, Casuccio A, Di Pace F, Morreale R, Pillitteri F, Cillino G, Lodato G. One-year outcomes with new-generation multifocal intraocular lenses. Ophthalmology. 2008 Sep;115(9):1508-16. doi: 10.1016/j.ophtha.2008.04.017. Epub 2008 Jun 5. PMID 18538402
- [Background] Cochener B; Concerto Study Group. Clinical outcomes of a new extended range of vision intraocular lens: International Multicenter Concerto Study. J Cataract Refract Surg. 2016 Sep;42(9):1268-1275. doi: 10.1016/j.jcrs.2016.06.033. PMID 27697244
- [Background] Davison JA, Simpson MJ. History and development of the apodized diffractive intraocular lens. J Cataract Refract Surg. 2006 May;32(5):849-58. doi: 10.1016/j.jcrs.2006.02.006. PMID 16765805
- [Background] de Silva SR, Evans JR, Kirthi V, Ziaei M, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2016 Dec 12;12(12):CD003169. doi: 10.1002/14651858.CD003169.pub4. PMID 27943250
- [Background] Harman FE, Maling S, Kampougeris G, Langan L, Khan I, Lee N, Bloom PA. Comparing the 1CU accommodative, multifocal, and monofocal intraocular lenses: a randomized trial. Ophthalmology. 2008 Jun;115(6):993-1001.e2. doi: 10.1016/j.ophtha.2007.08.042. Epub 2007 Nov 26. PMID 18031818
- [Background] Hashemi H, Khabazkhoob M, Soroush S, Shariati R, Miraftab M, Yekta A. The location of incision in cataract surgery and its impact on induced astigmatism. Curr Opin Ophthalmol. 2016 Jan;27(1):58-64. doi: 10.1097/ICU.0000000000000223. PMID 26569524
- [Background] Kaymak H, Hohn F, Breyer DR, Hagen P, Klabe K, Gerl RH, Mueller M, Auffarth GU, Gerl M, Kretz FT. [Functional Results 3 Months after Implantation of an "Extended Range of Vision" Intraocular Lens]. Klin Monbl Augenheilkd. 2016 Aug;233(8):923-7. doi: 10.1055/s-0042-104064. Epub 2016 Jul 6. German. PMID 27385257
- [Background] Lan J, Huang YS, Dai YH, Wu XM, Sun JJ, Xie LX. Visual performance with accommodating and multifocal intraocular lenses. Int J Ophthalmol. 2017 Feb 18;10(2):235-240. doi: 10.18240/ijo.2017.02.09. eCollection 2017. PMID 28251082
- [Background] Pedrotti E, Bruni E, Bonacci E, Badalamenti R, Mastropasqua R, Marchini G. Comparative Analysis of the Clinical Outcomes With a Monofocal and an Extended Range of Vision Intraocular Lens. J Refract Surg. 2016 Jul 1;32(7):436-42. doi: 10.3928/1081597X-20160428-06. PMID 27400074
- [Background] Prasher P, Sandhu JS. Prevalence of corneal astigmatism before cataract surgery in Indian population. Int Ophthalmol. 2017 Jun;37(3):683-689. doi: 10.1007/s10792-016-0327-z. Epub 2016 Aug 27. PMID 27567924
- [Background] TECNIS Symfony DFU
- [Background] Ruiz-Mesa R, Abengozar-Vela A, Aramburu A, Ruiz-Santos M. Comparison of visual outcomes after bilateral implantation of extended range of vision and trifocal intraocular lenses. Eur J Ophthalmol. 2017 Jun 26;27(4):460-465. doi: 10.5301/ejo.5000935. Epub 2017 Jan 28. PMID 28165609
- [Background] Weeber HA, Meijer ST, Piers PA. Extending the range of vision using diffractive intraocular lens technology. J Cataract Refract Surg. 2015 Dec;41(12):2746-54. doi: 10.1016/j.jcrs.2015.07.034. PMID 26796456
- [Result] Attia MSA, Auffarth GU, Kretz FTA, Tandogan T, Rabsilber TM, Holzer MP, Khoramnia R. Clinical Evaluation of an Extended Depth of Focus Intraocular Lens With the Salzburg Reading Desk. J Refract Surg. 2017 Oct 1;33(10):664-669. doi: 10.3928/1081597X-20170621-08. PMID 28991333
- [Result] Bellucci R. Multifocal intraocular lenses. Curr Opin Ophthalmol. 2005 Feb;16(1):33-7. doi: 10.1097/00055735-200502000-00006. PMID 15650577
- [Derived] Packer M, Monteiro T, Schweitzer C, Rosen P. Prospective, randomized, controlled multicenter study of a monofocal EDOF intraocular lens compared with a standard aspheric monofocal intraocular lens. J Cataract Refract Surg. 2025 Aug 1;51(8):659-665. doi: 10.1097/j.jcrs.0000000000001672. PMID 40245412